CLINICAL TRIAL: NCT03149302
Title: Effects of Local Neck Treatment With and Without Tailored Sensorimotor Control and Balance Exercises for Individuals With Chronic Neck Pain: Protocol for a Randomized Controlled Trial
Brief Title: Effects of Local Treatment With and Without Sensorimotor and Balance Exercises in Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chiang Mai University (Other)
Collaborators: The University of Queensland (Other); University of Applied Sciences and Arts of Southern Switzerland (Other)
Responsible Party: Principal Investigator, Sureeporn Uthaikhup, Principal Investigator, Chiang Mai University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: Chiangmai university
Record Dates: First submitted 2017-05-05; First posted 2017-05-11 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Neck Pain
Keywords: Manual therapy; Sensorimotor exercises; Balance exercises; Cervical mobilization; Specific neck muscle exercises
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Intervention Model Description: a 2 x 2 factorial blinded design
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Local neck treatment (LNT) (Experimental): Cervical mobilization and specific therapeutic exercises
  Interventions: Other: Local neck treatment (LNT)
- LNT plus sensorimotor exercises (Experimental): Local neck treatment plus a tailored sensorimotor exercise program.
  Interventions: Other: LNT plus sensorimotor exercises
- LNT plus balance exercises (Experimental): Local neck treatment plus balance training program.
  Interventions: Other: LNT plus balance exercises
- LNT plus sensorimotor/balance exercises (Experimental): A combination of local neck treatment, sensorimotor control exercise, and balance exercise.
  Interventions: Other: LNT plus sensorimotor/balance exercises

INTERVENTIONS:
Other: Local neck treatment (LNT) — The local neck treatment consists of cervical mobilization and specific therapeutic exercises (30 minutes). The participants will attend 12 individual treatment sessions (2 visits per week for 6 weeks).
  Arms: Local neck treatment (LNT)
Other: LNT plus sensorimotor exercises — The local neck treatment (30 minutes) plus the sensorimotor exercise program (15 minutes). The sensorimotor exercises include cervical joint position sense and oculomotor training. The participants will attend 12 individual treatment sessions (2 visits per week for 6 weeks).
  Arms: LNT plus sensorimotor exercises
Other: LNT plus balance exercises — The local neck treatment (30 minutes) plus the balance exercise program (15 minutes).The balance program includes with static balance and progress to dynamic balance and gait. The participants will attend 12 individual treatment sessions (2 visits per week for 6 weeks).
  Arms: LNT plus balance exercises
Other: LNT plus sensorimotor/balance exercises — The local neck treatment (30 minutes) plus the sensorimotor exercise program (15 minutes) and the balance exercises (15 minutes). The participants will attend 12 individual treatment sessions (2 visits per week for 6 weeks).
  Arms: LNT plus sensorimotor/balance exercises

SUMMARY:
The sensorimotor disturbance and postural instability have been demonstrated to be associated with neck pain. Specific therapeutic exercise and manual therapy for the cervical spine are effective interventions for improving dizziness symptoms, neck impairments, functional ability and quality of life. However, the effects of these interventions on the actual impairment of joint position sense and balance remain uncertain. Adaptive changes in the sensorimotor and postural control systems may need to be specifically addressed.

DETAILED DESCRIPTION:
The sensorimotor (joint position sense and oculomotor control) and postural stability (balance) disturbances have been demonstrated to be associated with neck pain. Specific therapeutic exercise directed to neuromuscular impairments and manual therapy for the cervical spine are effective interventions for improving dizziness symptoms, neck impairments, functional ability and quality of life. However, the effects of these interventions on the actual impairment of joint position sense and balance remain uncertain. Adaptive changes in the sensorimotor and postural control systems may need to be specifically addressed. Currently, it is not known whether the clinician has to train every impairment or can choose between sensorimotor training and balance training in the rehabilitation of neck pain. Different training approaches may have specific influences on the different outcomes and their outcomes will be important to inform the optimal and efficient management of persons with chronic neck pain.

ELIGIBILITY:
Inclusion Criteria:

* insidious neck pain for at least 3 months
* an average neck pain intensity over the past week ≥ 30 mm on a 100 mm visual analog scale (VAS)
* a score of neck pain and disability ≥ 10/ 100 on the Neck Disability Index-Thai version
* an absolute error of cervical joint position error > 4.5°
* an inability to stand in tandem stance with eyes closed for 30 seconds
* cervical segmental joint dysfunction (pain provoked >2/10 with abnormal tissue resistance)

Exclusion Criteria:

* a previous history of neck and head injury or surgery
* known or suspected vestibular pathology
* vertigo or dizziness caused by underlying pathology in the ear, brain, or sensory nerve pathways (e.g. benign paroxysmal positional vertigo and BPPV)
* vascular disorders (e.g. a migraine and hypertension)
* any musculoskeletal or neurological conditions that could affect a balance
* inflammatory joint disease
* systemic conditions
* cognitive impairment
* taking four or more medications
* received physiotherapy treatment for their neck disorder in the past 12 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-12-24 (Actual); Study Completion 2021-12-24 (Actual)

PRIMARY OUTCOMES:
Postural sway area | Change from baseline at immediate, and 3, 6, 12 months follow-ups
  The sway area during narrow stance on firm and soft surfaces with eyes open and eyes closed and during neck torsion maneuver (head turned 45 degrees to the left and right) on firm and soft surfaces, using a swaymeter device.
Postural sway displacement | Change from baseline at immediate, and 3, 6, 12 months follow-ups
  The sway displacement during narrow stance on firm and soft surfaces with eyes open and eyes closed and during neck torsion maneuver (head turned 45 degrees to the left and right) on firm and soft surfaces, using a swaymeter device.
Cervical joint position error | Change from baseline at immediate, and 3, 6, 12 months follow-ups
  The ability to perform an active movement (extension and rotation to the left and right) and return to the starting head position as accurately as possible, using a target on the wall and a laser-pointer attached to a lightweight headband.

SECONDARY OUTCOMES:
Gait speed | Change from baseline at immediate, and 3, 6, 12 months follow-ups
  Walk barefoot over 10 meters at a comfortable speed and then with head turns from side to side.
Dizziness intensity | Change from baseline at immediate, and 3, 6, 12 months follow-ups
  an average dizziness intensity over the past week on VAS 0-10
Neck pain intensity | Change from baseline at immediate, and 3, 6, 12 months follow-ups
  an average intensity of neck pain experienced in the past week on VAS 0-10.
Neck pain disability | Change from baseline at immediate, and 3, 6, 12 months follow-ups
  How neck pain affects a patient's daily life and to assess the self-rated disability, using NDI.
Pain extent | Change from baseline at immediate, and 3, 6, 12 months follow-ups
  Pain extent using a digital device (iPad Air 2) and sketching software (SketchBook Pro).
Pain location | Change from baseline at immediate, and 3, 6, 12 months follow-ups
  Pain location using a digital device (iPad Air 2) and sketching software (SketchBook Pro).
Cervical range of motion | Change from baseline at immediate, and 3, 6, 12 months follow-ups
  Cervical range of motion in flexion, extension, left-right lateral flexion and left-right rotation, using CROM.
Functional ability status | Change from baseline at immediate, and 3, 6, 12 months follow-ups
  Participants' functional status using the patient-specific functional scale (PSFS).
Health-related quality | Change from baseline at immediate, and 3, 6, 12 months follow-ups
  Participants' health-related quality of life, using Short Form-36.
Global perceived benefit of treatment | Change from baseline at immediate, and 3, 6, 12 months follow-ups
  Participant rated perceived benefit of treatment, using a six-point ordinal Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Sureeporn Uthaikhup, Ph.D., Principal Investigator — Department of physical therapy, Chiang Mai university
Locations (1):
- Department of Physical Therapy, Faculty of Associated Medical Sciences, Chiang Mai, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reid SA, Callister R, Katekar MG, Rivett DA. Effects of cervical spine manual therapy on range of motion, head repositioning, and balance in participants with cervicogenic dizziness: a randomized controlled trial. Arch Phys Med Rehabil. 2014 Sep;95(9):1603-12. doi: 10.1016/j.apmr.2014.04.009. Epub 2014 May 2. PMID 24792139
- [Background] Treleaven J, Peterson G, Ludvigsson ML, Kammerlind AS, Peolsson A. Balance, dizziness and proprioception in patients with chronic whiplash associated disorders complaining of dizziness: A prospective randomized study comparing three exercise programs. Man Ther. 2016 Apr;22:122-30. doi: 10.1016/j.math.2015.10.017. Epub 2015 Nov 26. PMID 26678652
- [Derived] Sremakaew M, Jull G, Treleaven J, Barbero M, Falla D, Uthaikhup S. Effects of local treatment with and without sensorimotor and balance exercise in individuals with neck pain: protocol for a randomized controlled trial. BMC Musculoskelet Disord. 2018 Feb 13;19(1):48. doi: 10.1186/s12891-018-1964-3. PMID 29433500